CLINICAL TRIAL: NCT04538937
Title: Prospective Registry of Eosinophilia With Respiratory Manifestations With Translational Research Identifying and Characterizing Eosinophils
Acronym: PROMETHEos
Status: Recruiting | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: 20200303-2218
Record Dates: First submitted 2020-08-25; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Eosinophilic Asthma; EGPA - Eosinophilic Granulomatosis With Polyangiitis; Samter Triad; HES - Hypereosinophilic Syndrome; Eosinophilic Pneumonia
MeSH Terms: conditions — Pulmonary Eosinophilia; Churg-Strauss Syndrome; Hypereosinophilic Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with eosinophilia and respiratory manifestation
  Interventions: Other: no intervention
- Healthy subjects
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Introduction: The etiology and therapy of eosinophilic lung diseases are still poorly understood. For individual forms of disease, such as eosinophilic asthma or eosinophilic granulomatosis with polyangiitis (EGPA), new therapeutic approaches exist that block the interleukin IL-5 or the IL-5 receptor. Eosinophilic manifestations of the respiratory tract can exclusively affect the lungs or occur as part of a systemic disease. The manifestations partially overlap and are clinically difficult to differentiate (e.g. eosinophilic asthma, Samter Triad, EGPA or hypereosinophilic syndrome (HES)). It is now known that blood eosinophil counts correlate with the level of eosinophils recruited to the airways. However, it is still unclear whether there is a blood eosinophilia without clinical relevance or whether there is a risk of organ damage (e.g. in HES). Hence, different subtypes of eosinophils with different polarization are discussed.

Aim of the study: A registry of patients with eosinophilia and respiratory manifestation will be established at the University Hospital of Innsbruck. The course of disease will be evaluated prospectively in a non-interventional study. This study stands on three main clinical pillars with focus on further characterization of eosinophilic cells:

1. Patients will be included who switch from a previous application of the anti-IL5 antibody mepolizumab (production and administration of the injection from lyophysate through the doctor) to the pre-mixed pen (self-injection at home).
2. Furthermore, special focus is set on patients suffering from the so-called Samter Triad. In these patients, the control of asthma, nasal polyps and NSAID intolerance will be examined in an interdisciplinary fashion during the course of treatment.
3. Previous clinical studies at our Department indicate that some patients with severe eosinophilic asthma or Samter Triad could represent a mono-organic or limited manifestation of lymphoid HES. This hypothesis is tested by measuring additional chemokines, somatic mutations and FACS parameters in this subgroup to verify a clonal disease.

In addition, translational research will differentiate resident and inflammatory eosinophilic granulocytes by FACS analysis and further characterize them by fluorescence microscopy, electron microscopy, gene chip analysis and lipidomics, in the above-mentioned diseases and in healthy controls, respectively.

Patients and methods: All patients suffering from eosinophilia with pulmonary involvement who are diagnosed with eosinophilic asthma, EGPA, Samter Triad, HES, and eosinophilic pneumonia with signed consent are included in the prospective registry. Provided, that they are registered at the outpatient department of pneumology, ENT, haematology or allergology at the University Hospital Innsbruck. The investigators will collect laboratory analyses, lung function, imaging, bone marrow biopsies, ENT findings and allergological findings over the course of the study. Furthermore, additional blood tubes are collected during routine blood tests, which are used to identify and characterize subtypes of eosinophilic granulocytes.

Risks for patients: No additional examinations, blood sampling or invasive measures are required for the patient. Thus, there is no additional risk for study participants.

Risks for control subjects: In order to be able to compare our results with the healthy population, volunteer subjects are recruited. After consent has been given, a blood sample is taken. Despite the low risk, it is theoretically possible that blood sampling may be accompanied by non-severe complications (such as hematoma, infection).

Benefits: The investigators expect new insights into phenotype and therapy of patients with eosinophilic manifestations of the respiratory tract.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* documented blood eosinophilia ≥ 300 cells/µl
* present tissue damage of the respiratory tract caused by eosinophils

Exclusion Criteria:

* age < 18 years
* pregnancy
* dementia
* incapacitated patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients suffering from severe, late-onset non-atopic eosinophilic asthma bronchiale on mepolizumab therapy or with planned mepolizumab therapy, recruited at our Dept. of Internal Medicine 2, Pneumology, Innsbruck Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-02-26 (Actual); Primary Completion 2021-02-26 (Estimated); Study Completion 2030-02-26 (Estimated)

PRIMARY OUTCOMES:
Establishment of a registry and descriptive characterization of the collective (frequencies of the individual types of disease, frequencies of the forms of therapy, documentation of the clinical course). | 10 years
Identification of inflammatory and regulatory eosinophils in peripheral blood by FACS analysis in all subtypes of eosinophilic manifestations of the respiratory tract | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic for Internal Medicine II, Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: No